CLINICAL TRIAL: NCT00812552
Title: Drug Eluting Stent Registry of Thrombosis
Acronym: DESERT
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DESERT
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Case: Late or very late drug-eluting stent thrombosis
- Control: No drug-eluting stent thrombosis

SUMMARY:
Multicenter, case-control study, to collect data regarding incidences of late and very late drug-eluting stent thrombosis with the aim of identifying trends and possible correlates of stent thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Case Subjects: patients who have experienced definite late or very late drug-eluting stent thrombosis
* Control Subjects: patients who underwent drug-eluting stent implantation at the same facility and in the same time period as a matched Case Subject, and have not experienced drug-eluting stent thrombosis.

Exclusion Criteria:

* Patients not meeting the above Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, male or female, over 18 years of age, who are either known to have experienced late or very late drug-eluting stent thrombosis (Case), or have undergone drug-eluting stent implantation at the same facility, in the same time period as a matched Case Subject, and have not experienced drug-eluting stent thrombosis (Control).
Sampling Method: Non-Probability Sample
Enrollment: 984 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To assess for potential correlates surrounding subjects and lesions among patients that experience late or very late drug-eluting stent thrombosis | Baseline

CONTACTS AND LOCATIONS:
Locations (20):
- United States (18):
  - Mercy General Hospital / Mercy Heart and Vascular Institute Cardiovascular Research, Sacramento, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Lexington Cardiac Research Foundation/Central Baptist Hospital, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Saint Luke's Hospital, Mid America Heart Institute, Kansas City, Missouri
  - The Valley Hospital, Ridgewood, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - Geisinger Health System, Danville, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - South Carolina Heart Center, PA, Columbia, South Carolina
  - Winchester Medical Center, Winchester, Virginia
- Laval Hospital, Québec, Quebec, Canada
- Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Waksman R, Kirtane AJ, Torguson R, Cohen DJ, Ryan T, Raber L, Applegate R, Waxman S, Gordon P, Kaneshige K, Leon MB; DESERT Investigators. Correlates and outcomes of late and very late drug-eluting stent thrombosis: results from DESERT (International Drug-Eluting Stent Event Registry of Thrombosis). JACC Cardiovasc Interv. 2014 Oct;7(10):1093-102. doi: 10.1016/j.jcin.2014.04.017. Epub 2014 Sep 17. PMID 25240540